CLINICAL TRIAL: NCT04926961
Title: Testing the Contribution of Orbitofrontal Cortex Networks to Reward Identity Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christina Zelano, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00214694
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Participants receive both sham TMS stimulation and real TMS stimulation in different sessions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham stimulation first, then real stimulation (Experimental): Participants will first be delivered sham TMS stimulation. Then on a separate day, participants will be delivered real TMS stimulation.
  Interventions: Device: Sham transcranial magnetic stimulation (TMS); Device: Real transcranial magnetic stimulation (TMS)
- Real stimulation first, then sham stimulation (Experimental): Participants will first be delivered real TMS stimulation. Then on a separate day, participants will be delivered sham TMS stimulation.
  Interventions: Device: Sham transcranial magnetic stimulation (TMS); Device: Real transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Sham transcranial magnetic stimulation (TMS) — Sham TMS will be applied using the MagVenture MagPro X100 stimulator with the placebo side of the Cool-B65 A/P coil.
Device: Real transcranial magnetic stimulation (TMS) — Real TMS will be applied using the MagVenture MagPro X100 stimulator with the active side of the Cool-B65 A/P coil.

SUMMARY:
This research study examines the contribution of orbitofrontal cortex (OFC) networks to learning reward identity expectations.

DETAILED DESCRIPTION:
This study is designed to examine the contribution of OFC networks to reward identity learning. It will use network-targeted TMS to test whether OFC is necessary for reward identity learning. Healthy human subjects will perform a three-reward reversal learning task after either TMS or sham stimulation while fMRI data are acquired. This is a randomized, within-subject, cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years old
* Right-handed
* Fluent English speakers

Exclusion Criteria:

* History of significant neurological conditions (e.g., epilepsy, dementia, multiple sclerosis, brain tumors, etc.)
* History of major psychiatric conditions (e.g., general anxiety disorder, depression, schizophrenia, obsessive-compulsive disorder, post-traumatic stress disorder, attention deficit hyperactivity disorder, alcoholism, etc.)
* Significant medical illnesses (e.g., cancer, meningitis, chronic obstructive pulmonary disease, cardiovascular disease, etc.)
* Significant cerebrovascular risk factors (e.g., hypertension, diabetes, elevated cholesterol, etc.)
* Current use of psychoactive medications (e.g., barbiturates, benzodiazepines, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, citalopram, escitalopram, fluoxetine, diazepam, etc.)
* Smell or taste dysfunction
* History of significant allergies requiring hospitalization for treatment
* History of severe asthma requiring hospitalization for treatment
* Habitual smoking
* Magnetic implants (e.g., shunts or stents, aneurysm clips, surgical clips, cochlear implants, metal bone/joint pins, plates and screws, eyelid spring or wires, etc.)
* Electronic devices (e.g., implanted cardiac defibrillator, cardiac pacemaker, deep brain/spinal cord or nerve stimulator, internal electrodes/wires, medication infusion devices, etc.)
* History of metal working without proper eye protection, or injury with metal shrapnel or metal slivers
* Claustrophobia
* Pregnancy
* Predisposition to seizures (e.g., personal history of seizures, family history of seizures epilepsy, pregnancy, alcoholism, etc.)
* Use of medications that increase the likelihood of seizures (e.g., bupropion, citalopram, duloxetine, ketamine, gamma-hydroxybutyrate, etc.)
* History of surgical procedures performed on the brain or spinal cord
* History of severe head trauma followed by loss of consciousness
* History of fainting spells or syncope
* Hearing problems or tinnitus

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

PRIMARY OUTCOMES:
Percentage of correct outcome predictions | 1 hour
  Percentage of correct outcome predictions in response to predictive cues during the reversal learning task.
Blood oxygen level-dependent (BOLD) responses | 1 hour
  Blood oxygen level-dependent (BOLD) responses measured using functional magnetic resonance imaging (fMRI) during the reversal learning task.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Zelano, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All data that underlie results in a publication
Time Frame: Upon publication
Access Criteria: Data can be obtained from PI for non-profit purposes upon reasonable request.